CLINICAL TRIAL: NCT00655603
Title: Influence of Glucagon Inhibition in Relation to the Anti-Diabetic Effect of GLP-1 in Patients With Type 2 Diabetes Mellitus.
Brief Title: Influence of Glucagon Inhibition in Relation to the Anti-Diabetic Effect of Glucagon-Like Peptide-1 (GLP-1) in Patients With Type 2 Diabetes Mellitus
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: University Hospital, Gentofte, Copenhagen (Other)
Collaborators: University of Copenhagen (Other); Hvidovre University Hospital (Other); Glostrup University Hospital, Copenhagen (Other)
Responsible Party: Kristine Juul Hare/MD, Gentofte University Hospital, Copenhagen
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Basic Science
Other Study IDs: H-C-2007-0072
Record Dates: First submitted 2008-04-04; First posted 2008-04-10 (Estimated); Last update posted 2009-04-06 (Estimated); Status verified 2009-04

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: GLP-1; Glucagon secretion; Glucose turn-over
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Glucagon-Like Peptide 1

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): 10 patients with Type 2 Diabetes Mellitus
  Interventions: Other: Infusion of native hormones from the pancreas and gut (GLP-1)
- 2 (Experimental): 10 healthy, matched control participants
  Interventions: Other: Infusion of native hormones from the pancreas and gut (GLP-1)

INTERVENTIONS:
Other: Infusion of native hormones from the pancreas and gut (GLP-1) — Glucose-clamps at fasting levels during infusion of hormones in different combinations.

SUMMARY:
Incretinbased treatment of patients with type 2 diabetes mellitus (T2DM) has increasing interest. The incretin glucagon-like peptide-1 (GLP-1) stimulates beta-cells to increased secretion and production of insulin. Glucose sensitivity is enhanced, apoptosis inhibited - progression in disease is potentially stopped. The alpha-cell is also influenced by GLP-1 as infusion lowers plasmaglucose (PG) levels in patients with type 1 diabetes mellitus (T1DM) (C-peptide negative) by inhibition of glucagon and thereby decreased hepatic glucoseproduction (HGP). Further Vilsboll et al has proved normalization of the glacgonostatic effect of glucose in patients with T2DM. As an attempt to elucidate glucose-intolerance in patients with T2DM further Knop et al investigated the glucagonresponse to both oral glucose tolerance test (OGTT) and a following iso-glycemic clamp. He saw a sufficient suppression of glucagon when glucose was introduced intravenously but the suppression of glucagon was attenuated and delayed when glucose was given orally.

The aim of this study is to elucidate the glucose intolerance further. Due to the complex interactions and mutual feed-back regulation between the pancreatic hormones and the PG level this protocol includes five days. All days include a euglycemic-clamp, patients with T2DM (n=10) are clamped at their fasting PG as are healthy control subjects (n=10). During the clamp either GLP-1 alone; GLP-1 in combination with somatostatin, insulin and glucagon; or somatostatin, insulin and glucagon are infused and blood samples are drawn.

The design of the study makes it possible to isolate the effect of each hormone. Further the investigators will be able to enlighten the effect of GLP-1 on the increase in glucose turn-over it induces.

The essential part in this design will be hormone concentrations and the response parameter the amount of glucose (AUC) it takes to create the euglycemic-clamp.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 Diabetes Mellitus according to criteria from WHO
* Normal hepatic and kidney function
* No overt diabetic complications
* Treatment with insulin or glitazones
* Informed consent

Exclusion Criteria:

* BMI < 23
* BMI > 35
* HbA1c > 10%
* Pregnancy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2008-03; Primary Completion 2009-05 (Estimated); Study Completion 2009-09 (Estimated)

PRIMARY OUTCOMES:
Glucose turn-over | 12 months

SECONDARY OUTCOMES:
The inhibitory effect of GLP-1 on glucagon, and the role of this in its anti-diabetic potential, measured by looking at glucose turn-over. | 12 months